CLINICAL TRIAL: NCT01515098
Title: The Effect of Blueberry Consumption on Cognition and Body Composition in Elderly Who Are Experiencing Mild Cognitive Decline
Brief Title: Effect of Blueberries on Cognition and Body Composition in Elderly With Mild Cognitive Decline
Acronym: BERRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Carol Cheatham, PhD, Assistant Professor of Psychology, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11-2075
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Mild Cognitive Decline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Blueberry Group (Experimental): 37 grams of dehydrated blueberries daily for 6 months
  Interventions: Dietary Supplement: Freeze-dried blueberries
- Placebo Group (Placebo Comparator): 37 grams of dextrose powder daily for 6 months
  Interventions: Dietary Supplement: Dextrose Placebo
- Reference Group (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Freeze-dried blueberries — Wild blueberries, freeze-dried and pulverized
  Arms: Blueberry Group
Dietary Supplement: Dextrose Placebo — Placebo developed to closely match blueberry powder.
  Arms: Placebo Group

SUMMARY:
Purpose: The purpose of this study is to examine the effect of blueberry consumption on cognitive decline and body composition in humans.

Hypothesis 1: Adults with mild cognitive decline who consume blueberries will experience an improvement in cognitive abilities as measured by a standardized battery of tests, relative to those who consume a placebo.

Hypothesis 2: Adults with mild cognitive decline who consume blueberries will evidence an increase in processing speed and an improvement in memory abilities as measured in an electrophysiological paradigm and compared to those who consume a placebo.

Hypothesis 3: Daily intake of 35 g freeze-dried blueberries will improve body composition (fat mass vs. lean mass).

Hypothesis 4: Daily intake of 35 g freeze-dried blueberries will decrease oxidative stress and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 65 and older
* BMI between 18.5 and 34.5
* Close individual to report memory decline

Exclusion Criteria:

* History of central nervous system or psychiatric disorders
* Dementia or Alzheimer's diagnosis
* Diabetes
* Smoking >20 cigarettes/day
* Gastrointestinal/digestive disorders
* Uncontrolled chronic disease

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in cognitive test performance | Baseline, 180 days
  Measured by CANTAB
Change in brain activity (N200, P300) related to cognitive abilities as measured by event-related potentials (ERP) | Baseline, 180 days
  Recognition memory, speed of processing, and memory consolidation as measured by the electrophysiological technique known as event-related potentials (ERP)

SECONDARY OUTCOMES:
Change in body mass distribution | Baseline, 180 days
  DXA scans to measure body composition at baseline and outcome will be compared for differences
Change in oxidative stress and inflammatory markers as measured in blood and urine | Baseline, 180 days
  Oxidative stress and inflammatory markers will be measured in blood and compared between baseline and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Cheatham, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Nutrition Research Institute, Kannapolis, North Carolina, United States

REFERENCES:
- [Derived] Cheatham CL, Canipe LG 3rd, Millsap G, Stegall JM, Chai SC, Sheppard KW, Lila MA. Six-month intervention with wild blueberries improved speed of processing in mild cognitive decline: a double-blind, placebo-controlled, randomized clinical trial. Nutr Neurosci. 2023 Oct;26(10):1019-1033. doi: 10.1080/1028415X.2022.2117475. Epub 2022 Sep 6. PMID 36066009
- [Derived] Sheppard KW, Cheatham CL. Omega-6/omega-3 fatty acid intake of children and older adults in the U.S.: dietary intake in comparison to current dietary recommendations and the Healthy Eating Index. Lipids Health Dis. 2018 Mar 9;17(1):43. doi: 10.1186/s12944-018-0693-9. PMID 29523147